CLINICAL TRIAL: NCT00276380
Title: A Phase III, Multicentre, Randomised, Double-blinded, Parallel Group, Placebo Controlled Clinical Study for Evaluating the Efficacy of EGb 761® (Tanakan®) (240mg) in the Recovery of Neurological Impairment Following Ischemic Stroke
Brief Title: A Study on the Use of Tanakan® for Recovery of Neurological Impairment Following Ischaemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-38-00240-704
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Stroke, Acute; Neurological Impairment
MeSH Terms: conditions — Stroke; Neurologic Manifestations | interventions — Ginkgo biloba extract; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGb761® (Experimental): EGb761® 240 milligrams (mg)/day for 6 months administered orally, in association with acetylsalicylic acid (325 mg/day).
  The test treatment consists of 6 tablets/day. 2 tablets (each containing 40 mg EGb761®) taken orally with half a glass of water during 3 main meals. 1 tablet/day of acetylsalicylic acid during lunch.
  Interventions: Drug: EGb761; Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): 6 months, administered orally, in association with acetylsalicylic acid (325 mg/day).
  The placebo consists of 6 tablets/day. 2 tablets taken orally with half a glass of water during 3 main meals. 1 tablet/day of acetylsalicylic acid during lunch.
  Interventions: Drug: Placebo; Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: EGb761 — EGb761 (Tanakan) 40 mg tablets (2 tablets t.i.d. (3 times a day)) 240 mg/day for 6 months.
  Other Names: Tanakan
  Arms: EGb761®
Drug: Placebo — Placebo 40 mg tablets (2 tablets t.i.d.) 240 mg/day for 6 months.
  Arms: Placebo
Drug: Acetylsalicylic acid — Acetylsalicylic acid 325 mg/day (1 tablet once daily), for 6 months.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Tanakan® 240mg in association with Acetylsalicylic acid (325mg/day) in the recovery of neurological impairment following ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient having had a single infarct in the carotid artery territory 3 to 8 days before inclusion
* Patient with a moderately severe or severe disability (Modified Rankin Score 4 or 5)
* Patient having a Quick's Test (for INR) and APPT (activated partial prothrombin time) test in the normal values of the laboratory

Exclusion Criteria:

* Patients having had an ischemic stroke (CT confirmed) less than 3 days and more than 8 days prior
* Patient with known pre-existent cerebral infarction
* Infarct damaged area bigger than 1/3 hemisphere
* Patient having a score below the cut-off point at Frenchay Aphasia Short Test

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2003-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- Czechia (2):
  - Faculty of Medicine in Hradec Kralove, Hradec Králové
  - General Faculty Hospital, Prague
- Poland (3):
  - Department and Clinic of Neurology of the Old Age, Katowice
  - CMUJ Krakov, Krakow
  - Postgraduate Medical Teaching Center, Warsaw
- Romania (2):
  - Institul de Boli Cerebro Vascular, Bucharest
  - Spitalul Universitar de Urgenta, Bucharest
- Russia (3):
  - Russian State Medical University - Neurology and Neurosurgery Clinic, Moscow
  - Russian State Medical University - Dept Fundamental Neurology & Neurosurgery, Moscow
  - Ural State Medical Academy, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre, international, randomised, double-blind, placebo-controlled study in which 204 subjects were enrolled in 8 centres, distributed in 4 countries: Romania, Poland, Czech Republic and Russian Federation, from 20 February 2003 to 25 February 2009.
Pre-assignment Details: The inclusion (baseline) visit on Day 0 was to take place within 3-8 days following an ischaemic stroke.
Groups:
- EGb761®: Subjects received EGb761® 240 milligrams (mg)/day for 6 months administered orally, in association with acetylsalicylic acid (325 mg/day).
  The test treatment consisted of 6 tablets/day. 2 tablets (each containing 40 mg EGb761®) were taken orally with half a glass of water during the 3 main meals. Subjects also took 1 tablet/day of acetylsalicylic acid during lunch.
- Placebo: Subjects received placebo for 6 months, administered orally, in association with acetylsalicylic acid (325 mg/day).
  The placebo consisted of 6 tablets/day. 2 tablets were taken orally with half a glass of water during the 3 main meals. Subjects also took 1 tablet/day of acetylsalicylic acid during lunch.
Period: Overall Study
Arm/Group | EGb761® | Placebo
Started | 102 | 102
Completed | 88 | 88
Not Completed | 14 | 14
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Death | 5 | 3
Not completed — Abnormal aPPT Levels | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- EGb761®: Subjects received EGb761® 240 mg/day for 6 months administered orally, in association with acetylsalicylic acid (325 mg/day).
  The test treatment consisted of 6 tablets/day. 2 tablets (each containing 40 mg EGb761®) were taken orally with half a glass of water during the 3 main meals. Subjects also took 1 tablet/day of acetylsalicylic acid during lunch.
- Total: Total of all reporting groups
Arm/Group | EGb761® | Placebo | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Median (Full Range); unit: years] | 68 [50 to 83] | 69 [50 to 90] | 68 [50 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 47 | 82
  Male | 67 | 55 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Modified Rankin Score of Less Than 3 at the End of Study Period.
Description: The degree of disability and dependence in daily activities was assessed using the modified Rankin scale. The modified Rankin scale is a 6-point numerical scale (0=no symptoms at all, 1=no significant disability, 2=slight disability, 3=moderate disability, 4=moderately severe disability, 5=severe disability) which measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168. The percentage of subjects having a modified Rankin Score<3 at the end of the study (Day 168) are reported.
Time Frame: Day 168
Population: This analysis was performed on the Intention-To-Treat (ITT) population which includes all subjects having at least one treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
percentage of participants | 59.8 | 64.7
Statistical Analysis 1: Comparison: EGb761® vs Placebo; The association between treatment and response after adjustment for the pooled centres was analysed using a Cochran-Mantel-Haenszel test; Test type: Other; p = 0.52, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.46 to 1.48] — The homogeneity of the Odds Ratio (OR) across centres was assessed by the Breslow Day test

2. Secondary Outcome: Percentage of Subjects With Modified Rankin Score of Less Than 3 at Day 28 and Day 84.
Description: The degree of disability and dependence in daily activities was assessed using the modified Rankin scale. The modified Rankin scale is a 6-point numerical scale (0=no symptoms at all, 1=no significant disability, 2=slight disability, 3=moderate disability, 4=moderately severe disability, 5=severe disability) which measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168. The percentage of subjects having a modified Rankin Score<3 at each follow-up visit (not including end of study) are reported.
Time Frame: Up to Day 84
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
percentage of participants
  Day 28 | 31.4 | 35.3
  Day 84 | 46.1 | 53.9
Statistical Analysis 1: Comparison: EGb761® vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Comparison of treatment effect at Day 28; p = 0.623, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.47 to 1.57] — The homogeneity of the Odds Ratio (OR) across centres was assessed by the Breslow Day test
Statistical Analysis 2: Comparison: EGb761® vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Comparison of treatment effect at Day 84; p = 0.3, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.42 to 1.3] — The homogeneity of the Odds Ratio (OR) across centres was assessed by the Breslow Day test

3. Secondary Outcome: Percentage of Subjects at Each Point on the Modified Rankin Scale at Baseline, Day 28, Day 84 and Day 168.
Description: The degree of disability and dependence in daily activities was assessed using the modified Rankin scale.The modified Rankin scale is a 6-point numerical scale (0=no symptoms at all, 1=no significant disability, 2=slight disability,3=moderate disability, 4=moderately severe disability, 5=severe disability) which measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168. The distribution of subjects according to disability severity scores was assessed and the percentage of subjects at each point on the modified Rankin scale are reported for each time point.
Time Frame: Up to Day 168
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
percentage of participants
  Day 0: No symptoms at all | 0 | 0
  Day 0: No significant disability | 0 | 0
  Day 0: Slight disability | 0 | 0
  Day 0: Moderate disability | 0 | 0
  Day 0: Moderately severe disability | 74.5 | 70.6
  Day 0: Severe disability | 25.5 | 29.4
  Day 28: No symptoms at all: number analyzed (Participants) | 97 | 96
  Day 28: No symptoms at all | 1.0 | 1.0
  Day 28: No significant disability: number analyzed (Participants) | 97 | 96
  Day 28: No significant disability | 7.2 | 9.4
  Day 28: Slight disability: number analyzed (Participants) | 97 | 96
  Day 28: Slight disability | 24.7 | 27.1
  Day 28: Moderate disability: number analyzed (Participants) | 97 | 96
  Day 28: Moderate disability | 38.1 | 31.3
  Day 28: Moderately severe disability: number analyzed (Participants) | 97 | 96
  Day 28: Moderately severe disability | 26.8 | 27.1
  Day 28: Severe disability: number analyzed (Participants) | 97 | 96
  Day 28: Severe disability | 2.1 | 4.2
  Day 84: No symptoms at all: number analyzed (Participants) | 93 | 89
  Day 84: No symptoms at all | 5.4 | 5.6
  Day 84: No significant disability: number analyzed (Participants) | 93 | 89
  Day 84: No significant disability | 24.7 | 25.8
  Day 84: Slight disability: number analyzed (Participants) | 93 | 89
  Day 84: Slight disability | 20.4 | 28.1
  Day 84: Moderate disability: number analyzed (Participants) | 93 | 89
  Day 84: Moderate disability | 38.7 | 27.0
  Day 84: Moderately severe disability: number analyzed (Participants) | 93 | 89
  Day 84: Moderately severe disability | 10.8 | 13.5
  Day 84: Severe disability: number analyzed (Participants) | 93 | 89
  Day 84: Severe disability | 0.0 | 0.0
  Day 168: No symptoms at all: number analyzed (Participants) | 88 | 88
  Day 168: No symptoms at all | 12.5 | 17.0
  Day 168: No significant disability: number analyzed (Participants) | 88 | 88
  Day 168: No significant disability | 29.5 | 31.8
  Day 168: Slight disability: number analyzed (Participants) | 88 | 88
  Day 168: Slight disability | 27.3 | 23.9
  Day 168: Moderate disability: number analyzed (Participants) | 88 | 88
  Day 168: Moderate disability | 25.0 | 20.5
  Day 168: Moderately severe disability: number analyzed (Participants) | 88 | 88
  Day 168: Moderately severe disability | 5.7 | 6.8
  Day 168: Severe disability: number analyzed (Participants) | 88 | 88
  Day 168: Severe disability | 0.0 | 0.0

4. Secondary Outcome: Mean Change From Baseline in Sandoz Clinical Assessment-Geriatric (SCAG) Scores at Day 28, Day 84 and Day 168.
Description: The SCAG scale was to be used to evaluate the psychopathological state of the subject. It is composed of 18 symptom areas and an overall global assessment, all rated on a 7-point format from 1=not present to 7=severe. The total score range is from 19 to 133 (best to worst), with a negative mean change from baseline indicating an improvement in symptoms. Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168 and the mean change from baseline at each time point is reported.
Time Frame: Up to Day 168
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
units on a scale
  Day 28: number analyzed (Participants) | 97 | 96
  Day 28 | -7.3 (5.9) | -5.0 (5.3)
  Day 84: number analyzed (Participants) | 93 | 89
  Day 84 | -8.8 (8.7) | -7.1 (6.6)
  Day 168: number analyzed (Participants) | 88 | 88
  Day 168 | -11.7 (8.2) | -9.2 (6.6)
Statistical Analysis 1: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 28; Test type: Other; p = 0.207, ANCOVA — Treatment effect was derived using a parametric analysis of covariance (ANCOVA) with baseline and pooled centres as covariates
Statistical Analysis 2: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 84; Test type: Other; p = 0.590, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates
Statistical Analysis 3: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 168; Test type: Other — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates; p = 0.814, ANCOVA

5. Secondary Outcome: Mean Change From Baseline in Barthel Index Scores at Day 28, Day 84 and Day 168.
Description: The performance in activities of daily living was assessed by using the Barthel scale. The Barthel scale is an ordinal scale which measures 10 performance items describing activities of daily living. Each item is rated with a given number of points from 0 indicating total dependence up to a maximum of 10 or 15 (depending on performance item) indicating complete independence. The total score range is from 0 to 100 (worst to best), with a positive mean change indicating an improvement in independence.
  Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168 and the mean change from baseline at each time point is reported.
Time Frame: Up to Day 168
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
units on a scale
  Day 28: number analyzed (Participants) | 97 | 96
  Day 28 | 31.2 (20.3) | 30.6 (18.6)
  Day 84: number analyzed (Participants) | 93 | 89
  Day 84 | 40.1 (19.9) | 41.5 (19.3)
  Day 168: number analyzed (Participants) | 88 | 88
  Day 168 | 46.3 (20.5) | 45.9 (19.2)
Statistical Analysis 1: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 28; Test type: Other; p = 0.240, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates
Statistical Analysis 2: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 84; Test type: Other; p = 0.441, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates
Statistical Analysis 3: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 168; Test type: Other; p = 0.645, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates

6. Secondary Outcome: Mean Change From Baseline in the Mini Mental State (MMS) Test Scores at Day 28, Day 84 and Day 168.
Description: The MMS test was used to evaluate the cognitive function of the subject. It includes tests of orientation, attention, memory, language and visual spatial skills, which are rated with a given number of points assigned to each level or ranking. The lower the score, the more important the mental deficit. The total score range is from 0 to 30 (worst to best), with a positive mean change indicating an improvement (i.e. less mental deficit). Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168 and the mean change from baseline at each time point is reported.
Time Frame: Up to Day 168
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
units on a scale
  Day 28: number analyzed (Participants) | 97 | 96
  Day 28 | 1.2 (1.9) | 1.2 (1.6)
  Day 84: number analyzed (Participants) | 93 | 89
  Day 84 | 1.4 (2.3) | 1.7 (2.3)
  Day 168: number analyzed (Participants) | 88 | 88
  Day 168 | 1.9 (2.7) | 2.0 (2.6)
Statistical Analysis 1: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 28; Test type: Other; p = 0.623, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates
Statistical Analysis 2: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 84; Test type: Other; p = 0.338, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates
Statistical Analysis 3: Comparison: EGb761® vs Placebo; Comparison of treatment effect at Day 168; Test type: Other; p = 0.828, ANCOVA — Treatment effect was derived using an ANCOVA analysis with baseline and pooled centres as covariates

7. Secondary Outcome: Mean Change From Baseline in the National Institute of Health Stroke Scale (NIHSS) Subscore for Questions 1a,1b and 1c at Day 28, Day 84 and Day 168.
Description: The NIHSS was to be used to objectively quantify the impairment caused by the stroke.The NIHSS is composed of 11 items, each of which score a specific ability between 0 (normal function) and 4 (high level of impairment).The minimum total score is 0 and maximum is 42. Only 8 of the NIHSS subscores were calculated for this study.
  Assessments were made at baseline (Day 0) and at each follow-up visit on Day 28, Day 84 and Day 168. Mean NIHSS subscores for questions 1a (level of consciousness),1b (asking patient the month and their age), and 1c (asking to open and close eyes) were analysed using descriptive quantitative statistics at each visit and the mean change from baseline at each time point is reported. The range for the subscore for items 1a is 0 - 3, for 1b is 0 - 2 and for 1c is 0 - 2 (best to worst), with a negative mean change from baseline indicating an improvement.
Time Frame: Up to Day 168
Population: This analysis was performed on the ITT population which includes all subjects having at least one treatment dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EGb761® | Placebo
Number analyzed (Participants) | 102 | 102
units on a scale
  Day 28: number analyzed (Participants) | 97 | 96
  Day 28 | -0.0 (0.2) | -0.0 (0.2)
  Day 84: number analyzed (Participants) | 93 | 89
  Day 84 | -0.0 (0.2) | -0.0 (0.1)
  Day 168: number analyzed (Participants) | 88 | 88
  Day 168 | -0.0 (0.2) | -0.0 (0.2)

ADVERSE EVENTS:
Time Frame: Up to Day 168
Description: All reported adverse events are treatment emergent adverse events (TEAEs). The analysis population is the Safety population which includes all subjects having received at least one treatment dose and one exploitable safety item after the instauration of treatment.
Arm/Group | EGb761® | Placebo
All-Cause Mortality (participants affected / at risk) | 5/101 | 3/100
Serious Adverse Events (participants affected / at risk) | 12/101 | 7/100
Other Adverse Events (participants affected / at risk) | 16/101 | 17/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGb761® (N=101) | Placebo (N=100)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) — AE had fatal outcome in 1 subject
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) — AE had fatal outcome
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — AE had fatal outcome
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) — AE had fatal outcome
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — AE had fatal outcome
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) — AE had fatal outcome
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — AE had fatal outcome
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — AE had fatal outcome
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) — AE had fatal outcome
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) — AE had fatal outcome
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGb761® (N=101) | Placebo (N=100)
Cystitis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No